CLINICAL TRIAL: NCT07158684
Title: Psychological Evaluation of Patients Undergoing Elective Surgery With Anxiety and Surgical Concerns: a Qualitative Interview Study
Brief Title: Surgical COrncerns and Psychological Evaluation of Patients Undergoing Elective Surgery
Acronym: SCOPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, Prof. Dr., University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 004382
Record Dates: First submitted 2025-07-11; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: Elective Surgery; Anxiety; Chronic Post Surgical Pain
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semi-structured interview (Experimental): A qualitative semi-structured interview of the patient's anxiety before and one month after surgery.
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — A qualitative semi-structured interview of the patient's anxiety before and one month after surgery.

SUMMARY:
This study wants to obtain more information regarding the patient's concerns since concerns of the patient about the procedure is found as a predictor for the development of chronic post-surgical pain. This step is crucial in translating early identification of a high-risk population into preventive policies. Using a semi-structured interview, the investigators aim to gather this additional information, which is essential in the development of an (individualized) biopsychosocial care pathway in the future.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Dutch speaking
* With a planned elective surgery, at the Antwerp University Hospital
* Score of ≥ 11 on APAIS anxiety subscale
* Must be able to complete questions on a tablet (digital literacy)
* Signed informed consen (prescreening informed consent and study participation informed consent)

Exclusion Criteria:

* Diagnostic procedures requiring anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Exploration of anxiety in patients undergoing elective surgery | before and one month after surgery
  Thematic analysis of the semi-structured interview response.

SECONDARY OUTCOMES:
To determine self-reported anxiety level regarding the surgical procedure before surgery. | From enrollment to pre-surgical visit
  by Amsterdam Preoperative Anxiety and Information Scale (APAIS) including six questionnaires (for anxiety and need for information). Scale ranging from 6-30. The higher the score the more anxiety and/or need for information.
To explore self-reported general depression level measured before surgery. | between pre-surgical visit and the day of surgery (Day 0)
  Beck Depression Inventory (BDI-2-NL)
To explore self-reported general anxiety level measured before surgery. | between pre-surgical visit and the day of surgery (Day 0)
  State-Trait Anxiety Inventory (STAI-Trait)
To explore self-reported moment-specific anxiety levels measured before and after surgery. | before surgery on the pre-surgical visit and 1 month after surgery
  by State-Trait Anxiety Inventory (STAI-State)
To explore pain intensity of the surgical site in patients before and after surgery | before surgery on the pre-surgical visit and 1 month after surgery
  by Numerical Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Antwerp, Edegem, Antwerpen, Belgium